CLINICAL TRIAL: NCT03423849
Title: Prospective Randomized Controlled Study of the Maintenance Regimen and Revised Regimen for Advanced Breast Cancer Survivors After First-line Salvage Therapy
Brief Title: The Maintenance Regimen and Revised Regimen for Advanced Breast Cancer Survivors After First-line Salvage Therapy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhiyong Yu (Other)
Responsible Party: Sponsor-Investigator, Zhiyong Yu, Director of the Breast Surgery Ⅰ, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShandongCHI-04
Record Dates: First submitted 2018-01-01; First posted 2018-02-06 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer; Chemotherapy Effect; Disease-free Survival
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine; Gemcitabine; Cisplatin; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The original program (NG/NP) (Experimental): Vinorelbine injection 25mg/m2 on day 1 and day 8, Gemcitabine injection 1250mg/m2 on day1 and day 8,every 3 weeks for 3 cycles（for the patients who used the NG salvage therapy） or Vinorelbine injection 25mg/m2 on day 1 and day 8,Cisplatin injection 25mg/m2 on day1,every 3 weeks for 3 cycles（for the patients who used the NP salvage therapy ）
  Interventions: Drug: Vinorelbine; Drug: Gemcitabine; Drug: Cisplatin
- One of the original program (N) (Experimental): Vinorelbine injection,25mg/m2 on day 1 and day 8,every 3 weeks for 6 cycles. or, Vinorelbine oral 60mg/m2 on day 1,every week for 6 cycles.
  Interventions: Drug: Vinorelbine
- Capecitabine monotherapy (Experimental): Capecitabine oral 1250mg/m2,bid,for 6 cycles
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Vinorelbine — 25mg/m2,day 1 and day 8, every 3 weeks
  Other Names: Anhydmvinblastine
  Arms: One of the original program (N); The original program (NG/NP)
Drug: Gemcitabine — 1250mg/m2,day 1 and day 8, every 3 weeks
  Other Names: Gemcel
  Arms: The original program (NG/NP)
Drug: Cisplatin — 25mg/m2,day 1,every 3 weeks
  Other Names: cisplatinum
  Arms: The original program (NG/NP)
Drug: Capecitabine — 1250mg/m2,day 1 to day 14, every 3 weeks
  Other Names: XELODA
  Arms: Capecitabine monotherapy

SUMMARY:
Worldwide, breast cancer is the most incident and prevalent cancer among women. Despite advances in the treatment of advanced breast cancer (ABC) during the past decade, adjuvant systemic therapy has yield little progression for such patients. ABC remains an incurable disease, responsible for approximate 40,000 deaths annually and a median life expectancy of no more than 3 years. The NCCN guidelines clearly define routine adjuvant chemotherapy regimens for the early breast cancer, however, for the patients with recurrence and metastasis, the choice of treatment options is not clear. In this trial, we choose the patients with disease progression who received anthracycline and taxane adjuvant chemotherapy after surgery. The patients received vinorelbine and gemcitabine (NG) or vinorelbine and platinum (NP) regiments for 6 cycles. Then the patients with complete response (CR), partly response (PR) and stable disease(SD) will be assigned to 3 groups, one group will receive the original regiment for 3 cycles to maintain treatment, one group will receive the vinorelbine for 6 cycles, the other group will receive the capecitabine for 6 cycles. Trasuzumab will be used to patients if HER-2 positive. Endocrine therapy will be used if the hormone receptors positive after the chemotherapy. The primary endpoint is to assess disease-free survival (DFS), the secondary endpoint is to assess the overall survival (OS).

DETAILED DESCRIPTION:
The trial is designed to help us to choose the maintain treatment regiment for the patients with effective first-line salvage therapy. After inorelbine and gemcitabine (NG) or vinorelbine and platinum (NP) regiments for 6 cycles, patients will be assess the effect of treatment. As for the patients with complete response (CR), partly response (PR) and stable disease(SD), the investigators will randomly assign them to receive 3 cycles of original regiment, or 6 cycles of vinorelbine, or 6 cycles of capecitabine. Trasuzumab will be used to patients if HER-2 positive. Endocrine therapy will be used if the hormone receptors positive after the chemotherapy. The effectiveness of therapy will be estimated after the maintain therapy. The first two years the patient was prescribed every 3 months to review the disease, then review the disease every six months. The primary endpoint is to assess disease-free survival (DFS), the secondary endpoint is to assess the overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* All patients were required to give written informed consent.
* Patients with distant metastasis who primary received anthracycline and taxane adjuvant chemotherapy after surgery.
* After inorelbine and gemcitabine (NG) or vinorelbine and platinum (NP) regiments for 6 cycles,patients were assessed the effect of treatment. As for the patients with complete response (CR), partly response (PR) and stable disease(SD).
* Have normal cardiac functions by echocardiography
* ECOG scores are ≤ 0-1.
* Patients are disposed to practice contraception during the whole trial.
* The results of patients' blood tests are as follows:

Hb ≥ 90 g/L WBC ≥ 3.0×109/L Plt ≥ 100×109/L Neutrophils ≥ 1.5×109/L ALT and AST ≤ 2.5 times of normal upper limit. TBIL ≤ 1.5 times of normal upper limit. Creatinine ≤ 1.5 times of normal upper limit.

Exclusion Criteria:

* Have other cancers at the same time or have the history of other cancers in recent five years, excluding the controlled skin basal cell carcinoma or skin squamous cell carcinoma or carcinoma in situ of cervix.
* Active infections.
* Severe non-cancerous diseases.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-02-08 (Estimated); Primary Completion 2020-02-08 (Estimated); Study Completion 2020-02-08 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 5 years
  To determine the percentage of disease-free survival (DFS) for the The original program (NG/NP) or One of the original program (N) or Capecitabine monotherapy

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  To determine the percentage of Overall survival (OS) for the The original program (NG/NP) or One of the original program (N) or Capecitabine monotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyong Yu, PhD, Study Chair — Shandong Cancer Hospital and Institute; Zhaoyun Liu, MD, Principal Investigator — Shandong Cancer Hospital and Institute